CLINICAL TRIAL: NCT01101009
Title: Efficacy of Sevikar® Compared to the Combination of Perindopril/ Amlodipine on Central Arterial Blood Pressure in Patients With Moderate to Severe Hypertension-
Brief Title: Comparison of Sevikar® and the Combination of Perindopril/Amlodipine on Central Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSE- SEV-02-09; 2009-012966-30 (EudraCT Number)
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2013-01

CONDITIONS: Hypertension
Keywords: Sevikar®; Central Arterial Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Perindopril; Amlodipine; Hydrochlorothiazide; olmesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perindopril+amlodipine (Active Comparator)
  Interventions: Drug: Perindopril + amlodipine + if necessary, hydrochlorothiazide
- Olmesartan/amlodipine (Active Comparator)
  Interventions: Drug: olmesartan/amlodipine + hydrochlorothiazide, if necessary.

INTERVENTIONS:
Drug: Perindopril + amlodipine + if necessary, hydrochlorothiazide — Two perindopril 4 mg tablets + 1 amlodipine 10 mg tablet + placebo tablet matching the olmesartan/amlodipine tablet. All tablets are taken once daily. The duration of administration of perindopril tablets and placebo is 24 weeks. The duration of administration of amlodipine tablets is 24-26 weeks. Hydrochlorthiazide tablets 12.5 mg or 25 mg, once daily, will be added, if necessary
  Arms: Perindopril+amlodipine
Drug: olmesartan/amlodipine + hydrochlorothiazide, if necessary. — olmesartan/amlodipine tablets 40 mg/10 mg, + placebo tablets matching the perindopril tablet and amlodipine tablet. All tablets are taken once daily for 24 weeks. Hydrochlorthiazide tablets 12.5 mg or 25 mg, once daily, will be added, if necessary
  Arms: Olmesartan/amlodipine

SUMMARY:
Comparison of the combination of amlodipine with an angiotensin receptor blocker or an angiotensin converting inhibitor, on central arterial blood pressure in patients with hypertension and additional risk factors. This is a randomised, double-blind, double-dummy, multicenter study. The duration of active treatment 24 weeks.

DETAILED DESCRIPTION:
The study, multi-center balanced, parallel group (two treatment arms), randomized, double-blind (double-dummy), non-inferiority study is designed to show non-inferiority of Sevikar® (olmesartan(OM)/amlodipine (AM)) 40/10 mg compared to the combination of Perindopril (PER) 8 mg plus Amlodipine 10 mg with regard to central systolic blood pressure lowering effect, using the change from baseline (Week 0) to final examination (Week 24).

Male and female Caucasians aged ≥ 40 years and <80 years with moderate to severe hypertension, defined by a systolic blood pressure (SBP) ≥ 160 and ≤ 200 or diastolic blood pressure (DBP) ≥ 100 and ≤ 115 mmHg for untreated patients, SBP ≥ 140 or DBP ≥ 90 mmHg for insufficiently pre-treated patients and SBP ≥ 130 mmHg or DBP ≥ 80 mmHg for insufficiently pretreated diabetics chronic kidney disease will be eligible for participation. In addition,three additional risk factors should be present.

During the course of the study three central blood pressure measurements (at randomization, at week 12 and at termination) will be performed with SphygmoCor ultrasound method. The conventional measurements with calibrated tensiometers (Omron) will be performed at each visit. Ambulatory blood pressure monitoring will be performed at randomisation.

The study starts with a 2-4 week run in phase. AM will be given as open-labelled 5 mg or 10 mg tablets, administered once daily. After randomization during the double-blind phase, study medication will comprise either OM/AM 40/10 mg or PER 8 mg (2x4 mg) plus AM 10 mg and will be administered once daily. Furthermore, open-label HCTZ 12.5 mg and 25.0 mg will be provided in tablets and administered once daily according to the treatment schedule.

The primary endpoint is the change in central SBP from baseline (Week 0, Visit 0) to final examination (Week 24, Visit 5) using Last Observation Carried Forward (LOCF) approach.

The study is conducted in approximately 15 centres in Spain. Depending on the previously administered drugs the run in phase is up to four weeks (Visits -2 and -1). Individual duration of active treatment (after randomization) will last 24 weeks (Visits 0-5). The total individual duration is 28 weeks.

A total of 518 patients (259 patients/arm) will be needed in the Per Protocol Set (PPS) for the confirmatory primary analysis using mean change from baseline (Week 0) to Final Examination assuming a drop out rate of 20% during Run-in Phase a total of 720 patients have to be screened in order to achieve 576 (288 patients/arm) randomised patients.

Assuming approximately 10% major protocol deviations, a total of 518 patients will remain in the PPS.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe hypertension
* 3 additional risk factors such as age > 55 (male), > 65 female, smoker, type 2 diabetes, obesity, cardiovascular disease, congestive heart failure, chronic kidney disease,
* ability to give informed consent

Exclusion Criteria:

* secondary or malignant hypertension
* contraindication to any of the study drugs
* Creatinine clearance level <40ml/min
* treatment with more than 3 antihypertensive drugs
* Myocardial infarction, percutaneous transluminal coronary angioplasty, cardiac bypass surgery < 6 month prior to start of the study,
* unstable angina pectoris,
* stroke, transient ischemic attack < 3 months prior to start,
* Congestive heart failure NYHA II-IV,
* clinically relevant concomitant diseases,
* alcohol or drug abuse,
* pregnancy or women of childbearing potential without contraceptive precaution,

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in central systolic blood pressure from baseline (Week 0, Visit 0) to Final Examination (Week 24, Visit 5) using last observation carried forward approach. | Baseline to week 24

SECONDARY OUTCOMES:
Changes in systolic and diastolic ambulatory blood pressure (mean of 24h, daytime and night-time) | Baseline to week 24
Changes in conventional mean sitting systolic and diastolic blood pressure measurement | Baseline to 24 weeks
Incidence and profile of AEs separately by Run-in Phase and by double-blind Treatment Phase | Run in phase (2 weeks) to end of study (24 weeks)
Number of responders at Final Examination defined as normalized or a decrease of systolic blood pressure by at least 20 mmHg or diastolic blood pressure by at least 10 mmHg in conventional BP measurements. | Baseline to 24 weeks
Number of normalized at Final Examination (defined as blood pressure <140/90 mmHg or <130/80 mmHg in diabetics/chronic kidney disease, in conventional BP measurements. | Baseline to 24 weeks
Changes in mean sitting systolic and diastolic blood pressure (BP) measurements from week 12 to Final Exam in patients with stabilized BP (BP is < 140/90 mmHg or < 130/80 mmHg for diabetics/chronic kidney disease) from Week 12 and Week 18. | Week 12 to Week 18 or week 24
Changes in Central Systolic Blood Pressure from week 12 to Final Examination in patients with stabilised BP (i.e. patients whose BP is < 140/90 mmHg or < 130/80 mmHg for diabetics/chronic kidney disease) between Week 12 and Week 18. | Week 12 to week 18 or week 24

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Centro de Salud Casas Ibañez, Albacete
  - Hospital del Mar, Barcelona
  - Hospital General de Jerez de la Frontera, Cadiz
  - Hospital Universitario de Fuenlabrada, Fuenlabrada (Madrid)
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital General Universitario La Paz, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario de Móstoles, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Carlos Haya, Málaga
  - Centro de Salud Murcia San Andrés, Murcia
  - Hospital de Sagunto, Puerto de Sagunto (Valencia)
  - Centro de Salud La Alamedilla, Salamanca
  - Hospital Virgen de la Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Ruilope L, Schaefer A. The fixed-dose combination of olmesartan/amlodipine was superior in central aortic blood pressure reduction compared with perindopril/amlodipine: a randomized, double-blind trial in patients with hypertension. Adv Ther. 2013 Dec;30(12):1086-99. doi: 10.1007/s12325-013-0076-6. Epub 2013 Nov 30. PMID 24293132
- [Derived] Ruilope LM, Schaefer A. Efficacy of Sevikar(R) compared to the combination of perindopril plus amlodipine on central arterial blood pressure in patients with moderate-to-severe hypertension: Rationale and design of the SEVITENSION study. Contemp Clin Trials. 2011 Sep;32(5):710-6. doi: 10.1016/j.cct.2011.04.011. Epub 2011 May 14. PMID 21586342